CLINICAL TRIAL: NCT01205607
Title: IRB-HSR# 14299: The Use of the Intrathoracic Pressure Regulator (ITPR) to Improve Cerebral Perfusion Pressure in Patients With Altered Intracranial Elastance
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Virginia (Other)
Responsible Party: Edward C., Nemergut MD, University of Virginia Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 14299
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ITPR -9 & then -5 mm Hg (Experimental): the ITPR will be inserted in the ventilator circuit and activated to provide either -5 mm Hg or -9 mm Hg endotracheal tube pressure (ETP) Each subject will have all measurements recorded at both -5 & -9 mm Hg
  Interventions: Device: ITPR -9 & then -5mm Hg
- ITPR -5 & then _9 mm HG (Experimental): the ITPR will be inserted in the ventilator circuit and activated to provide either -5 mm Hg or -9 mm Hg endotracheal tube pressure (ETP) Each subject will have all measurements recorded at both -5 & -9 mm Hg
  Interventions: Device: ITPR -5 mm Hg then -9 mm Hg

INTERVENTIONS:
Device: ITPR -5 mm Hg then -9 mm Hg — the ITPR will be inserted in the ventilator circuit and activated to provide either -5 mm Hg or -9 mm Hg endotracheal tube pressure (ETP) Each subject will have all measurements recorded at both -5 & -9 mm Hg
  Arms: ITPR -5 & then _9 mm HG
Device: ITPR -9 & then -5mm Hg — the ITPR will be inserted in the ventilator circuit and activated to provide either -5 mm Hg or -9 mm Hg endotracheal tube pressure (ETP) Each subject will have all measurements recorded at both -5 & -9 mm Hg
  Arms: ITPR -9 & then -5 mm Hg

SUMMARY:
Patients who have a functioning intracranial pressure-monitoring device (either a subarachnoid bolt, or an intraventricular catheter) in place, and are either sedated, intubated, and mechanically ventilated (i.e. in the NNICU), or are scheduled to undergo an operation or interventional neuroradiological procedure at the University of Virginia. Patients with a contraindication to TTE will be excluded.

For patients in the NNICU, basic hemodynamic variables (systemic blood pressure, central venous pressure, etc.) will be collected. In addition, left ventricular performance (including estimates of LVEDV, LVESV, EF, FAC, and SV) will be assessed using TTE. Once these baseline data are recorded, the ITPR will be inserted in the ventilator circuit and activated to provide either -5 mm Hg or -9 mm Hg endotracheal rube pressure (ETP) (based on a randomization scheme). After the ITPR has been active for at least five minutes, the same intracranial, hemodynamic, and TTE data obtained above will be gathered. The ITPR will then be turned off for five minutes, and intracranial, hemodynamic, and TTE data will again be recorded. The ITPR will be activated a second time (-9 mm Hg or -5 mm Hg ETP, i.e. whichever value was not used previously), and after five minutes of use data will be recorded again. The ITPR will then be disconnected, data will be collected after waiting two minutes, and no further interventions will be made.

ABG's will be obtained before and during the use of the device at each setting.

This is a proof of concept/feasibility study designed to test the primary hypothesis that use of the ITPR will result in decreased intracranial pressure and increased cerebral perfusion pressure. The effect of the ITPR on secondary indicators of cardiac performance will also be examined. These include but are not limited estimates of ventricular end diastolic volume and pressure (LVEDV/P), ejection fraction (EF), left ventricular end systolic volume and pressure (LVESV/P), fractional area change (FAC), all of which will be assessed by transthoracic echocardiography (TTE) or transesophageal echocardiography (TEE).

DETAILED DESCRIPTION:
The ITPR is an FDA-approved device intended to increase circulation and blood pressure in hypovolemic and cardiogenic shock. The device is inserted within a standard respiratory circuit between the patient and the ventilator. It functions by decreasing intrathoracic pressure during the expiratory phase to subatmospheric levels after each positive pressure ventilation. This decrease in intrathoracic pressure creates a vacuum within the thorax relative to the rest of the body, thereby enhancing venous return to the heart and consequently increasing cardiac output and blood pressure. Activation of the device is also accompanied by a decrease in SVR. The end result is a device that simultaneously improves cardiac output by increasing LVEDV and decreasing SVR while increasing coronary perfusion pressure by increasing blood pressure and decreasing LVESP/LVESV.1-8

Interestingly, while the ITPR was developed as a non-invasive mechanism to increase preload in hypovolemic patients, its mechanism of action (generation of subatmospheric intrathoracic pressure) has been shown to reduce intracranial pressure6. This is critical in brain-injured patients, because elevated intracranial pressure is strongly associated with poor outcome in traumatic brain injury (TBI) patients - in a recent study of 846 TBI patients, those with ICP < 20 mm Hg by 48 hours had a mortality rate of 14%, whereas those with ICP > 20 mm Hg had a mortality rate of 34%9. Particularly interesting are the ITPR's combined benefits of increased MAP and decreased ICP, as hypotension is a well-known poor prognostic indicator in this patient population.

In fact, according to the Brain Trauma Foundation Guidelines, "Hypotension, occurring at any time from injury through the acute intensive care course, has been found to be a primary predictor of outcome from severe head injury for the health care delivery systems within which prognostic variables have been best studied. Hypotension is repeatedly found to be one of the five most powerful predictors of outcome and is generally the only one of these five that is amenable to therapeutic modification. A single recording of a hypotensive episode is generally associated with a doubling of mortality and a marked increase in morbidity from a given head injury10."

Importantly, cerebral perfusion pressure (mean arterial pressure - the greater of ICP or CVP) is only a surrogate marker for cerebral blood flow. The function of hypotension as a useful clinical variable is dependent on two factors - first, its correlation with the true variable of interest (cerebral blood flow) and second, the ability of clinicians to manipulate the underlying variable of interest (cerebral blood flow) based on the surrogate marker (cerebral perfusion pressure).

The acceptable level of hypotension in patients with brain injuries has not been determined, and the Brain Trauma Foundation (BTF) Guidelines recommend maintaining systolic blood pressures > 90 mm Hg, but acknowledge that this number is relatively arbitrary and not based on any high-level studies (thus assigning it a designation of Level II evidence) 11. The BTF Guidelines further state that because hypotension is such a poor prognostic variable, it would be unethical to randomize patients to various blood pressure goals, and therefore Level I evidence is not forthcoming. Further complicating the situation is the lack of agreement on how to increase blood pressure (with the hopes of increasing cerebral perfusion pressure)12-15. Many of the pharmacologic agents used to increase mean arterial pressure have significant vasoconstrictive effects, which could counteract any increase blood pressure and lead to unchanged, or even reduced cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

* 1. patients who have a functioning intracranial pressure-monitoring device (either a subarachnoid bolt, or an intraventricular catheter) in place, and are either sedated, intubated, and mechanically ventilated (i.e. in the NNICU)and have an arterial line in place, or are scheduled to undergo an operation or interventional neuroradiological procedure at the University of Virginia.

  2. age 18 years of age and older 3. informed consent/ surrogate consent has been obtained

Exclusion Criteria:

* 1. pneumothorax 2. hemothroax 3. uncontrolled bleeding 4. uncontrolled hypertension defined as SBP > 180 mmHg at the time of surgery 5. known respiratory disease such as chronic emphysema, COPD, or Cystic Fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
Hemodynamic variables | baseline, 5 minutes after device activation & 5 minutes after device turned off
  hemodynamic variables (systemic blood pressure, central venous pressure, ICP) will be collected at baseline, 5 minutes after device activation & 5 minutes after device turned off

SECONDARY OUTCOMES:
cardiac performance | baseline, 5 minutes after device activation & 5 minutes after device turned off
  cardiac performance will also be examined. These include but are not limited estimates of ventricular end diastolic volume and pressure (LVEDV/P), ejection fraction (EF), left ventricular end systolic volume and pressure (LVESV/P), fractional area change (FAC)

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Nemergfut, MD, Principal Investigator — University of Virginia Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Lurie KG, Zielinski TM, McKnite SH, Idris AH, Yannopoulos D, Raedler CM, Sigurdsson G, Benditt DG, Voelckel WG. Treatment of hypotension in pigs with an inspiratory impedance threshold device: a feasibility study. Crit Care Med. 2004 Jul;32(7):1555-62. doi: 10.1097/01.ccm.0000131207.29081.a2. PMID 15241102
- [Background] Lurie KG, Zielinski T, McKnite S, Aufderheide T, Voelckel W. Use of an inspiratory impedance valve improves neurologically intact survival in a porcine model of ventricular fibrillation. Circulation. 2002 Jan 1;105(1):124-9. doi: 10.1161/hc0102.101391. PMID 11772887
- [Background] Lurie KG, Voelckel WG, Zielinski T, McKnite S, Lindstrom P, Peterson C, Wenzel V, Lindner KH, Samniah N, Benditt D. Improving standard cardiopulmonary resuscitation with an inspiratory impedance threshold valve in a porcine model of cardiac arrest. Anesth Analg. 2001 Sep;93(3):649-55. doi: 10.1097/00000539-200109000-00024. PMID 11524335
- [Background] Lurie KG, Mulligan KA, McKnite S, Detloff B, Lindstrom P, Lindner KH. Optimizing standard cardiopulmonary resuscitation with an inspiratory impedance threshold valve. Chest. 1998 Apr;113(4):1084-90. doi: 10.1378/chest.113.4.1084. PMID 9554651
- [Background] Yannopoulos D, McKnite S, Metzger A, Lurie KG. Intrathoracic pressure regulation improves 24-hour survival in a porcine model of hypovolemic shock. Anesth Analg. 2007 Jan;104(1):157-62. doi: 10.1213/01.ane.0000249047.80184.5a. PMID 17179262
- [Background] Yannopoulos D, McKnite SH, Metzger A, Lurie KG. Intrathoracic pressure regulation for intracranial pressure management in normovolemic and hypovolemic pigs. Crit Care Med. 2006 Dec;34(12 Suppl):S495-500. doi: 10.1097/01.CCM.0000246082.10422.7E. PMID 17114984
- [Background] Yannopoulos D, Metzger A, McKnite S, Nadkarni V, Aufderheide TP, Idris A, Dries D, Benditt DG, Lurie KG. Intrathoracic pressure regulation improves vital organ perfusion pressures in normovolemic and hypovolemic pigs. Resuscitation. 2006 Sep;70(3):445-53. doi: 10.1016/j.resuscitation.2006.02.005. Epub 2006 Aug 9. PMID 16901611
- [Background] Yannopoulos D, Nadkarni VM, McKnite SH, Rao A, Kruger K, Metzger A, Benditt DG, Lurie KG. Intrathoracic pressure regulator during continuous-chest-compression advanced cardiac resuscitation improves vital organ perfusion pressures in a porcine model of cardiac arrest. Circulation. 2005 Aug 9;112(6):803-11. doi: 10.1161/CIRCULATIONAHA.105.541508. Epub 2005 Aug 1. PMID 16061732
- [Background] Jiang JY, Gao GY, Li WP, Yu MK, Zhu C. Early indicators of prognosis in 846 cases of severe traumatic brain injury. J Neurotrauma. 2002 Jul;19(7):869-74. doi: 10.1089/08977150260190456. PMID 12184856
- [Background] The Brain Trauma Foundation. The American Association of Neurological Surgeons. The Joint Section on Neurotrauma and Critical Care. Hypotension. J Neurotrauma. 2000 Jun-Jul;17(6-7):591-5. doi: 10.1089/neu.2000.17.591. PMID 10937905
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. I. Blood pressure and oxygenation. J Neurotrauma. 2007;24 Suppl 1:S7-13. doi: 10.1089/neu.2007.9995. No abstract available. PMID 17511549
- [Background] Pfister D, Strebel SP, Steiner LA. Effects of catecholamines on cerebral blood vessels in patients with traumatic brain injury. Eur J Anaesthesiol Suppl. 2008;42:98-103. doi: 10.1017/S0265021507003407. PMID 18289425
- [Background] Dudkiewicz M, Proctor KG. Tissue oxygenation during management of cerebral perfusion pressure with phenylephrine or vasopressin. Crit Care Med. 2008 Sep;36(9):2641-50. doi: 10.1097/CCM.0b013e3181847af3. PMID 18679110
- [Background] Myburgh JA. Driving cerebral perfusion pressure with pressors: how, which, when? Crit Care Resusc. 2005 Sep;7(3):200-5. PMID 16545046
- [Background] Alspaugh DM, Sartorelli K, Shackford SR, Okum EJ, Buckingham S, Osler T. Prehospital resuscitation with phenylephrine in uncontrolled hemorrhagic shock and brain injury. J Trauma. 2000 May;48(5):851-63; discussion 863-4. doi: 10.1097/00005373-200005000-00008. PMID 10823528